CLINICAL TRIAL: NCT01569828
Title: An Open Label, Parallel-group Study to Determine Multiple Dose Pharmacokinetics of LCZ696 and Its Metabolites in Subjects With Severe Renal Impairment Compared to Matched Healthy Subjects With Normal Renal Function
Brief Title: Multiple Dose Pharmacokinetics of LCZ696 and Its Metabolites in Subjects With Severe Renal Impairment vs. Matched Healthy Subjects With Normal Renal Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLCZ696A2205; 2007-005482-36
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Results first posted 2015-09-29 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-08

CONDITIONS: Pharmacokinetics; Renal Impaired; Healthy Volunteer
Keywords: LCZ696; pharmacokinetics

ARMS (2):
- Renal Impaired Subjects (Experimental): once daily administration of 400 mg LCZ696 for 5 days
  Interventions: Drug: LCZ696A
- Healthy Volunteers (Experimental): once daily administration of 400 mg LCZ696 for 5 days
  Interventions: Drug: LCZ696A

INTERVENTIONS:
Drug: LCZ696A
  Arms: Renal Impaired Subjects
Drug: LCZ696A — once daily administration of 400 mg LCZ696 for 5 days
  Arms: Healthy Volunteers

SUMMARY:
An open label, parallel-group study to determine multiple dose pharmacokinetics of LCZ696 and its metabolites in subjects with severe renal impairment compared to matched healthy subjects with normal renal function

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Novartis Investigative Site, Neuss, Germany
- Novartis Investigative Site, Moscow, Russia
- Novartis Investigative Site, Belgrade, Serbia

RESULTS

PARTICIPANT FLOW:
Groups:
- Severe Renal Impaired Subjects: Subjects with severe (CrCl from <30 mL/min), renal function who were otherwise in good health as determined by past medical history, physical examination, electrocardiogram, vital signs (measured after 3 minutes rest in the supine position) which are within the following ranges; oral body temperature between 35.0-37.8°C, systolic blood pressure (95-180 mm Hg), diastolic blood pressure (60-110 mm Hg), pulse rate (54-95 bpm), laboratory tests and urinalysis. Creatinine clearance (CrCl) was calculated by the Cockcroft-Gault (CG) formula with patient stratification based on the screening serum creatinine measurement. Once daily administration of 400 mg LCZ696 p.o. for 5 days
- Matched Healthy Volunteers: All healthy volunteers were matched by age (±5 years), sex and BMI (±10%) to the renal subjects enrolled into the study. Subjects were to be in good health as determined by past medical history, physical examination, electrocardiogram, vital signs (measured after 3 minutes rest in the supine position) which are within the following ranges; oral body temperature between 35.0-37.2 °C, systolic blood pressure (95-140 mm Hg), diastolic blood, pressure (60-100 mm Hg), pulse rate (45-90 bpm), laboratory tests and urinalysis. Healthy subjects must have a CrCl of >80 mL/min.Once daily administration of 400 mg LCZ696 p.o. for 5 days
Period: Overall Study
Arm/Group | Severe Renal Impaired Subjects | Matched Healthy Volunteers
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Matched Healthy Volunteers: All healthy volunteers were matched by age (±5 years), sex and BMI (±10%) to the renal subjects enrolled into the study. Subjects were to be in good health as determined by past medical history, physical examination, electrocardiogram, vital signs (measured after 3 minutes rest in the supine position) which are within the following ranges; oral body temperature between 35.0-37.2 °C, systolic blood pressure (95-140 mm Hg), diastolic blood, pressure (60-100 mm Hg), pulse rate (45-90 bpm), laboratory tests and urinalysis. Healthy subjects must have a CrCl of >80 mL/min.
  Once daily administration of 400 mg LCZ696 p.o. for 5 days
- Total: Total of all reporting groups
Arm/Group | Severe Renal Impaired Subjects | Matched Healthy Volunteers | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (7.76) | 52.5 (6.98) | 53.2 (7.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Time to Reach Maximum Peak Plasma Concentration (Tmax) After Single Dose (Day 1), and After Multiple Dose Administration (Day 5)
Time Frame: 1 and 5 days
Population: Pharmacokinetic analysis set
Measure: Median (Full Range); unit: hour
Groups:
- Renal Impaired Subjects: Subjects with severe (CrCl from <30 mL/min), renal function who were otherwise in good health as determined by past medical history, physical examination, electrocardiogram, vital signs (measured after 3 minutes rest in the supine position) which are within the following ranges; oral body temperature between 35.0-37.8°C, systolic blood pressure (95-180 mm Hg), diastolic blood pressure (60-110 mm Hg), pulse rate (54-95 bpm), laboratory tests and urinalysis. Creatinine clearance (CrCl) was calculated by the Cockcroft-Gault (CG) formula with patient stratification based on the screening serum creatinine measurement. Once daily administration of 400 mg LCZ696 p.o. for 5 days
- Healthy Volunteers: All healthy volunteers were matched by age (±5 years), sex and BMI (±10%) to the renal subjects enrolled into the study. Subjects were to be in good health as determined by past medical history, physical examination, electrocardiogram, vital signs (measured after 3 minutes rest in the supine position) which are within the following ranges; oral body temperature between 35.0-37.2 °C, systolic blood pressure (95-140 mm Hg), diastolic blood, pressure (60-100 mm Hg), pulse rate (45-90 bpm), laboratory tests and urinalysis. Healthy subjects must have a CrCl of >80 mL/min. Once daily administration of 400 mg LCZ696 p.o. for 5 days
Arm/Group | Renal Impaired Subjects | Healthy Volunteers
Number analyzed (Participants) | 6 | 6
hour
  AHU377 (Sacubitril) on day 1 | 0.5 [0.5 to 1] | 0.5 [0.5 to 1.0]
  AHU377 (Sacubitril) on day 5 | 0.5 [0.5 to 1.0] | 0.5 [0.5 to 0.5]
  LBQ657(Sacubitril pro-drug) on day 1 | 3 [2 to 4] | 3 [2 to 4]
  LBQ657(Sacubitril pro-drug) on day 5 | 2 [2 to 4] | 2.5 [2 to 4]
  VAL489 (valsartan) on day 1 | 2 [1 to 3] | 2 [2 to 2]
  VAL489 (valsartan) on day 5 | 2 [1 to 3] | 2 [1 to 2]

2. Secondary Outcome: 24 hr Sodium Urinary Excretion in Subjects With Severe Renal Impairment and Their Matched Healthy Volunteers
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: mmol/day
Arm/Group | Renal Impaired Subjects | Healthy Volunteers
Number analyzed (Participants) | 6 | 6
mmol/day
  baseline | 172.658 (79.9239) | 177.833 (39.5533)
  Day 1 | 133.000 (35.5564) | 187.000 (42.8392)
  Day 2 | 89.333 (34.5714) | 156.833 (26.4607)
  Day 3 | 106.050 (39.6424) | 145.500 (31.5325)
  Day 4 | 94.683 (21.3792) | 140.500 (30.9629)
  Day 5 | 93.500 (36.2171) | 156.667 (32.1165)
  Day 6 | 88.400 (23.1383) | 96.167 (28.6316)
  Day 7 | 107.150 (36.1899) | 107.667 (57.4514)

3. Primary Outcome: (Cmax) After Single Dose (Day 1), and After Multiple Dose Administration (Day 5)
Time Frame: 1 and 5 days
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Renal Impaired Subjects | Healthy Volunteers
Number analyzed (Participants) | 6 | 6
ng/mL
  AHU377 (Sacubitril)on day 1 | 5215 (3220) | 2810 (862)
  AHU377(Sacubitril) on day 5 | 4960 (3430) | 2407 (1780)
  LBQ657 (Sacubitril prodrug)on day 1 | 15967 (3380) | 14633 (2233)
  LBQ657 ( Sacubitril prodrug) on day 5 | 30650 (11462) | 18233 (1975)
  VAL489 (valsartan) on day 1 | 5935 (2191) | 4988 (1093)
  VAL489 (valsartan) on day 5 | 5852 (3306) | 5672 (1314)

4. Primary Outcome: AUC 0-24h After Single Dose (Day 1), and After Multiple Dose Administration (Day 5)
Time Frame: 1 and 5 days
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: (hr*ng/mL)
Arm/Group | Renal Impaired Subjects | Healthy Volunteers
Number analyzed (Participants) | 6 | 6
(hr*ng/mL)
  AHU377 (Sacubitril) on day 1 | 5918 (3430.4) | 4101 (815.36)
  AHU377(Sacubitril) on day 5 | 5495 (2890.2) | 4336 (745.88)
  LBQ657(Sacubitril prodrug) on day 1 | 254000 (72562) | 146100 (17346)
  LBQ657 (Sacubitril prodrug) on day 5 | 538300 (268650) | 185500 (29759)
  VAL489 (valsartan) on day 1 | 40560 (11344) | 29870 (8756.9)
  VAL489 (valsartan) on day 5 | 51080 (33780) | 32470 (8687.1)

5. Primary Outcome: T1/2 After Multiple Dose Administration (Day 5)
Description: Summary statistics for plasma PK parameters following 5 days QD dose of 400mg LCZ696
Time Frame: 5 days
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: (hr)
Arm/Group | Renal Impaired Subjects | Healthy Volunteers
Number analyzed (Participants) | 6 | 6
(hr)
  AHU377 (Sacubitril)on day 5 | 2.030 (1.2793) | 1.916 (0.69234)
  LBQ657(Sacubitril prodrug) on day 5 | 38.55 (17.301) | 13.16 (2.6829)
  VAL489 (valsartan) on day 5 | 26.40 (9.1992) | 12.98 (2.9882)

6. Primary Outcome: CL/F After Multiple Dose Administration (Day 5)
Description: Summary statistics for plasma PK parameters following 5 days QD dose of 400mg LCZ696
Time Frame: 5 days
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: (ml/hr)
Arm/Group | Renal Impaired Subjects | Healthy Volunteers
Number analyzed (Participants) | 6 | 6
(ml/hr)
  AHU377(Sacubitril) on day 5 | 45100 (24523) | 45900 (8168.0)
  LBQ657( Sacubitril prodrug) on day 5 | NA (NA) — LBQ657 is a metabolite of AHU377, and hence LBQ657 CL/F values are not relevant. | NA (NA) — LBQ657 is a metabolite of AHU377, and hence LBQ657 CL/F values are not relevant.
  VAL489 (valsartan) on day 5 | 7370 (8063.0) | 6792 (2051.1)

7. Primary Outcome: CLr After Multiple Dose Administration (Day 5)
Description: Summary statistics for plasma PK parameters following 5 days QD dose of 400mg LCZ696
Time Frame: 5 days
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: (ml/hr)
Groups:
- Renal Impaired Subjects: Subjects with severe (CrCl from <30 mL/min), renal function who were otherwise in good health as determined by past medical history, physical examination, electrocardiogram, vital signs (measured after 3 minutes rest in the supine position) which are within the following ranges; oral body temperature between 35.0-37.8°C, systolic blood pressure (95-180 mm Hg), diastolic blood pressure (60-110 mm Hg), pulse rate (54-95 bpm), laboratory tests and urinalysis. Creatinine clearance (CrCl) was calculated by the Cockcroft-Gault (CG) formula with patient stratification based on the screening serum creatinine measurement.Once daily administration of 400 mg LCZ696 p.o. for 5 days
Arm/Group | Renal Impaired Subjects | Healthy Volunteers
Number analyzed (Participants) | 6 | 6
(ml/hr)
  AHU377 (Sacubitril) on day 5 | 24.18 (28.781) | 111.8 (82.310)
  LBQ657 (Sacubitril prodrug) on day 5 | 47.39 (38.392) | 436.9 (72.388)
  VAL489 (valsartan) on day 5 | 28.89 (20.781) | 299.4 (97.887)

ADVERSE EVENTS:
Time Frame: Serious Adverse Events are monitored from date of First Subject First Visit (FSFV) until Last Subject Last Visit (LSLV). All other adverse events are monitored from First Subject First Treatment (FSFT) until Last Subject Last Visit (LSLV).
Arm/Group | Severe Renal Impaired Patients | Matched Healthy Volunteers
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Severe Renal Impaired Patients (N=6) | Matched Healthy Volunteers (N=6)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 3 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Somnolence (Nervous system disorders) | 0 | 1
Diastolic hypertension (Vascular disorders) | 1 | 0
Orthostatic hypertension (Vascular disorders) | 3 | 0
Orthostatic hypotension (Vascular disorders) | 3 | 0
Systolic hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial